CLINICAL TRIAL: NCT02694081
Title: The Advantages and Disadvantages Between Uncut Roux-en-Y Reconstruction
Brief Title: The Advantages and Disadvantages Between Uncut Roux-en-Y Reconstruction and Billroth II Reconstruction After Laparoscopy-assisted Distal Gastrectomy for Gastric
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Aiping shi, Assisted Investigator, Jilin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 130021; 714488468 (Other: Department of Gastrointestinal and Anal Surgery)
Record Dates: First submitted 2016-01-29; First posted 2016-02-29 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-07

CONDITIONS: Gastric Cancer
Keywords: reflux; residue; Gastric stasis; Emptying time
MeSH Terms: conditions — Stomach Neoplasms; Gastroesophageal Reflux; Gastroparesis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Uncut Roux-en-Y Reconstruction (Experimental): Uncut Roux-en-Y Reconstruction will be used after laparoscopy-assisted distal gastrectomy for early gastric cancer.
  Interventions: Procedure: Uncut Roux-en-Y Reconstruction
- Billroth II Reconstruction (Active Comparator): Billroth II Reconstruction will be used after laparoscopy-assisted distal gastrectomy for early gastric cancer.
  Interventions: Procedure: Billroth II Reconstruction

INTERVENTIONS:
Procedure: Uncut Roux-en-Y Reconstruction — All surgical procedures will be performed by the single surgery team ,which is leaded by professor Wang Quan. Uncut Roux-en-Y construction will be used in this group.
  Arms: Uncut Roux-en-Y Reconstruction
Procedure: Billroth II Reconstruction — All surgical procedures will be performed by the single surgery team ,which is leaded by professor Wang Quan. Uncut Roux-en-Y construction will be used in this group.
  Arms: Billroth II Reconstruction

SUMMARY:
The Advantages and Disadvantages Between Uncut Roux-en-Y Reconstruction and Billroth II Reconstruction After Laparoscopy-assisted Distal Gastrectomy for Gastric.

DETAILED DESCRIPTION:
To search which is the better reconstructions by comparing and analyzing the advantages and disadvantages between Uncut Roux-en-Y and Billroth II reconstructions after laparoscopy-assisted distal gastrectomy for gastric cancer.

Method: It's a prospective study including all patients underwent laparoscopy-assisted distal gastrectomy (LADG) in the First Hospital of Jilin University, from February 2016 to February 2017. All surgical procedures will be performed by the single surgery team, which is leaded by professor Wang Quan. The reconstruction method will be selected randomly from Uncut Roux-en-Y and Billroth II anastomosis by drawing lots preoperatively without distinct indications. Clinical data, operation data and perioperative complications and related physiological indexes of differences.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of distal gastric cancer
* underwent laparoscopy-assisted distal gastrectomy

Exclusion Criteria:

* have simultaneously other cancer
* have severe systemic inflammatory disease ,serious illness such as diabetes, chronic lung diseases
* have upper gastrointestinal surgery
* can't bear the gastric tube
* the period is too late or the tumor is too large to carry on a laparoscopy assisted radical distal gastrectomy

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
The time of reconstruction during operations of Uncut Roux-en-Y Reconstruction and Billroth II Reconstruction | within 2 hours after surgery
  The time of reconstruction operation will be recorded in the operating note by nurses in minutes.
change of potential of hydrogen ( pH) in remnant stomach | 1-6 days after surgery
  In the morning of 1-6 days after operation , monitor the number of gastric juice's potential of hydrogen ( pH) value through gastric tube and write down the data. So if the data is greater than 7,the complication of bile reflux happened
the amount of blood loss during operations of Uncut Roux-en-Y Reconstruction and Billroth II Reconstruction | within 2 hours after surgery
  During the operation the amount of blood loss will be recorded in the operating note by nurses in milliliters.

SECONDARY OUTCOMES:
the number of patients with the complication of Residual food | 6 month after surgery
  During the upper gastrointestinal radiography，if there is residual food,the meglumine diatrizoate will be separate and then write down the number.
the number of patients with the complication of Reflux esophagitis | 6 month after surgery
  During the upper gastrointestinal radiography,if there is meglumine diatrizoate refluxing to esophagus,it will be observed and written down in number.

OTHER OUTCOMES:
the number of patients with the complication of gastroesophageal reflux disease(GERD) | 6 month after surgery
  all patients of this clinical trial will be investigated by Gastroesophageal reflux disease questionnaire(GerdQ),and all patients whose score is beyond 8 will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Wang, professor, Study Director — The First Hospital of Jilin University
Locations (1):
- the first hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Cai Z, Mu M, Ma Q, Liu C, Jiang Z, Liu B, Ji G, Zhang B. Uncut Roux-en-Y reconstruction after distal gastrectomy for gastric cancer. Cochrane Database Syst Rev. 2024 Feb 29;2(2):CD015014. doi: 10.1002/14651858.CD015014.pub2. PMID 38421211